CLINICAL TRIAL: NCT05091424
Title: A Phase IB Open-Label, Multicenter Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Mosunetuzumab and a Combined Regimen of Mosunetuzumab and Venetoclax in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Brief Title: A Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Mosunetuzumab and a Combined Regimen of Mosunetuzumab and Venetoclax in Participants With Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO43243
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — tocilizumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Participants with R/R CLL who have failed two prior lines of therapy and who have had prior exposure to BTKi and/or venetoclax will receive mosunetuzumab subcutaneous (SC) monotherapy
  Interventions: Drug: Mosunetuzumab; Drug: Tocilizumab
- Arm B (Experimental): Participants with R/R CLL who have failed two prior lines of therapy, who are currently progressing on BTKi therapy, and who require salvage therapy as assessed by their treating physician will receive mosunetuzumab SC with BTKi overlap therapy for the first two cycles of mosunetuzumab SC
  Interventions: Drug: Mosunetuzumab; Drug: Tocilizumab
- Arm C (non-US participants only) (Experimental): Participants with R/R CLL who have failed two prior lines of therapy and who have had prior exposure to BTKi and/or venetoclax will receive mosunetuzumab SC with venetoclax (this arm is open only to participants outside of the US)
  Interventions: Drug: Mosunetuzumab; Drug: Tocilizumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Mosunetuzumab — Participants will receive subcutaneous (SC) mosunetuzumab
  Other Names: Lunsumio
Drug: Tocilizumab — Participants will receive intravenous (IV) tocilizumab as needed for cytokine release syndrome (CRS) events.
Drug: Venetoclax — Participants will receive daily oral venetoclax
  Other Names: Venclyxto; Venclexta
  Arms: Arm C (non-US participants only)

SUMMARY:
This study will assess the safety, tolerability, pharmaokinetics, and preliminary efficacy of mosunetuzumab (Lunsumio) monotherapy in participants with relapsed or refractory (R/R) chronic lymphocytic leukemia (CLL). This study will also allow participants who are currently progressing on a Bruton tyrosine kinase inhibitor (BTKi) and requiring salvage therapy as assessed by the treating physician to continue their BTKi throughout the screening period and for the first two cycles of mosunetuzumab. An additional arm (open to non-US participants only) has been added to assess the safety, tolerability, pharmacokinetics, and preliminary efficacy of mosunetuzumab in combination with venetoclax, a B-cell lymphoma 2 (BCL2) inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of CLL requiring treatment according to the International Workshop on CLL (iwCLL) criteria (Hallek et al 2018)
* Eastern Cooperative Oncology Group (ECOG) performance score (PS) of ≤ 2
* Adequate bone marrow (BM) function independent of growth factor or transfusion support, within 2 weeks of screening, at screening as defined by the protocol unless cytopenia is clearly due to marrow involvement of CLL
* Adequate liver function unless directly attributable to the participant's CLL
* Life expectancy > 6 months
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year, and agreement to refrain from donating eggs during the treatment period and for at least 3 months after the last dose of mosunetuzumab and 3 months after the last dose of tocilizumab (if applicable)
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm as defined by the protocol

Inclusion Criteria Specific to Arm B:

* Participants must have been taking a BTKi for at least 12 months, have demonstrated evidence of progressive disease while receiving the BTKi and require additional salvage therapy as assessed by their treating physician. Participants should be able to continue their previously prescribed BTKi at a stable dose throughout the study screening period and for the first two cycles of mosunetuzumab administration

Inclusion Criteria Specific to Arm C:

* Non-US participants only

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of mosunetuzumab and tocilizumab or within 30 days after the final dose of venetoclax (if applicable)
* Participants who have received any of the following treatments prior to study entry: treatment with mosunetuzumab or other CD20/CD3-directed bispecific antibodies; allogenic stem cell transplant
* Participants who have received any of the following treatments, whether investigational or approved, within the respective time periods prior to initiation of study treatment: radiotherapy within 2 weeks prior to the first dose of study treatment; autologous stem cell transplant within 100 days prior to first study treatment; CAR T-cell therapy within 30 days before first study treatment; prior use of any monoclonal antibodies, radioimmunoconjugates, or antibody-drug conjugates for anti-CLL treatment within 4 weeks before first dose of study treatment; systemic immunosuppressive medications (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to the first dose of study treatment; any other anti-cancer therapy, whether investigational or approved, including but not limited to chemotherapy within 4 weeks prior to initiation of study treatment (except for participants enrolled in Arm B, where overlapping therapy is permitted; other prior cancer immunotherapy not explicitly defined by the protocol is to be discussed with the medical monitor to determine eligibility
* Received a live, attenuated vaccine within 4 weeks before the first dose of study treatment, or in whom it is anticipated that such a vaccine will be required during the study period or within 5 months after the final dose of study treatment
* Transformation of CLL to aggressive non-Hodgkin's lymphoma (NHL)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* Contraindication to tocilizumab
* History of prior malignancy except for conditions defined by the protocol
* Participants with infections requiring intravenous (IV) treatment with antibiotics or hospitalization within the last 4 weeks prior to enrollment or known active bacterial, viral (including SARS-CoV-2), fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment
* Evidence of any significant concomitant disease that could affect compliance with the protocol or interpretation of results
* Recent major surgery within 4 weeks prior to first study treatment administration, with the exception of protocol-mandated procedures (e.g., tumor biopsies and bone marrow biopsies)
* Positive SARS-CoV-2 test within 7 days prior to enrollment

Exclusion Criteria Specific to Arm C:

* Have received venetoclax therapy within 12 months prior to first study treatment administration
* Participants with known infection with HIV or human T-cell leukemia virus 1 (HTLV1)
* HIV testing will be performed in countries where mandatory testing by health authorities is required
* HTLV testing is required in participants from endemic countries
* Participants with uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia
* Participants who have received the following: strong and moderate CYP3A inhibitors within 7 days prior to the initiation of study treatment; strong and moderate CYP3A inducers within 7 days prior to the initiation of study treatment; steroid therapy for anti-neoplastic intent with the exception of inhaled steroids for asthma, topical steroids, or replacement/stress corticosteroids within 7 days prior to the first dose of study drug administration
* Have consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit within 3 days prior to the first dose of study drug and throughout venetoclax administration
* Inability to swallow a large number of tablets
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Known allergy to both xanthine oxidase inhibitors and rasburicase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of Dose-Limiting Toxicities (DLTs) | Up to approximately 12 months (Arms A and B) or 24 months (Arm C)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 8-12 weeks after the last dose of study drug
Minimal Residual Disease (MRD) Response Rate | Up to 8-12 weeks after the last dose of study drug
Progression-Free Survival (PFS) | From the first study treatment to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 12 months (Arms A and B) or 24 months (Arm C))
Overall Survival (OS) | From the first dose of study drug to death from any cause (up to approximately 12 months (Arms A and B) or 24 months (Arm C))
Event-Free Survival (EFS) | Between the date of the first study treatment to the date of disease progression/relapse, death, or start of new anti-leukemic therapy, whichever occurs first (up to approximately 12 months (Arms A and B) or 24 months (Arm C))
Complete Response (CR) Rate | Up to 8-12 weeks after the last dose of study drug
Duration of Response (DOR) | From the first occurrence of a documented objective response to disease progression by iwCLL 2018 criteria or death from any cause (up to approximately 12 months (Arms A and B) or 24 months (Arm C))
Percentage of Participants with Adverse Events (AEs) | Up to approximately 12 months (Arms A and B) or 24 months (Arm C)
Maximum Serum Concentration (Cmax) of Mosunetuzumab SC | Up to approximately 12 months (Arms A and B) or 24 months (Arm C)
Minimum Serum Concentration (Cmin) of Mosunetuzumab SC | Up to approximately 12 months (Arms A and B) or 24 months (Arm C)
Time to Maximum Concentration (Tmax) of Mosunetuzumab SC | Up to approximately 12 months (Arms A and B) or 24 months (Arm C)
Incidence of Anti-Drug Antibodies (ADAs) | Baseline through end of study (up to approximately 12 months for Arms A and B, or 24 months for Arm C)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (31):
- United States (5):
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Uni of Texas - Md Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute at The University of Utah, Salt Lake City, Utah
- Australia (3):
  - Princess Alexandra Hospital Woolloongabba, Woolloongabba, Queensland
  - Peter MacCallum Cancer Center, East Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
- China (4):
  - Peking University People's Hospital, Beijing
  - Southern Medical University Nanfang Hospital, Guangzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Tianjin Institute of Hematology & Blood Diseases Hospital, Tianjin
- France (2):
  - Chu de Clermont Ferrand, Clermont-Ferrand
  - IUCT Oncopole, Toulouse
- Germany (3):
  - Universitätsklinikum Augsburg, Augsburg
  - Uniklinik Koln, Cologne
  - Universitätsklinikum Ulm, Ulm
- Italy (4):
  - A.O. Spedali Civili Di Brescia-P.O. Spedali Civili, Brescia, Lombardy
  - Osp. San Raffaele, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia, Sant'Andrea Delle Fratte (PG), Umbria
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - PRATIA MCM Kraków, Krakow
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroc?aw
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Yeouido St. Mary's Hospital, Seoul
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
- United Kingdom (2):
  - Christie Hospital NHS Trust, Manchester
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No